CLINICAL TRIAL: NCT05002426
Title: Rouviere Sulcus Plane and Hepatic Hilum Plane, Which is Better as a Landmark in Laparoscopic Bile Duct Surgerys
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Second Hospital of Anhui Medical University (Other)
Responsible Party: Principal Investigator, hui hou, The Second Hospital of Anhui Medical University, The Second Hospital of Anhui Medical University
Other Study IDs: 1458
Record Dates: First submitted 2021-08-04; First posted 2021-08-12 (Actual); Last update posted 2021-08-12 (Actual); Status verified 2021-08

CONDITIONS: Cholelithiasis; Laparoscopic Cholecystectomy
Keywords: anatomy
MeSH Terms: conditions — Cholelithiasis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- The type and orientation of Rouviere sulcus: "open type", "fused type" or "absent type"

SUMMARY:
RS and the RS plane are important anatomical markers in laparoscopic cholecystectomy. However, there are many variations in the shape and orientation of the RS, and the RS plane is an imaginary plane, which can be misjudged by different surgeons. The purpose of this study is to introduce a more intuitive anatomical marker and anatomical plane, hilum plane, and discuss the application value of hilum plane in laparoscopic biliary surgery by comparing it with RS and RS plane.

DETAILED DESCRIPTION:
Hepatic hilum plane is the hepatoduodenal serosa plane that extends from the base of the liver IVa segment down to the first segment of the gallbladder triangle.

During the operation, first pulling the gallbladder to the head side, using the separating forceps to slide down horizontally from the hilum (the basement of hepatic segment Ⅳ), and along the serous of hepatoduodenal ligament, that is so called "hilum plane".

It forms a "neck-shoulder" structure when the hilar plane meets the tent-like hepatobiliary triangle. the serosa of hepatobiliary triangle was dissected on the neck area and ventral side of hilar plane, and the serosa of posterior triangle of the gallbladder was also cutted on the same extension line . In this process, the type and orientation of RS, the relationship between the plane of the RS sulcus and the plane of the hilar plane were also recorded and compared with hilum plane.

ELIGIBILITY:
Inclusion Criteria:

Benign disease of the gallbladder requires surgery

Exclusion Criteria:

Patients with severe cirrhosis or had a history of partial hepatectomy were excluded from the statistics .

patients with unexpected gallbladder carcinoma.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: a consecutive patients undergoing elective laparoscopic cholecystectomies at the second affiliated hospital of Anhui medical university
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-01-04 (Actual); Primary Completion 2021-10-01 (Estimated); Study Completion 2021-10-01 (Estimated)

PRIMARY OUTCOMES:
The type of Rouviere sulcus and the "fake RS" | up to 30 days after surgery
  The Rouviere sulcus was present if a fissure was seen in the liver parenchyma on the right side of the gallbladder and continues with the right posterior hepatic pedicle(fig ). RS were further subdivided into three classes: "open type", "fused type" or "absent type"). The "plane of RS sulcus" was also recorded If the RS was not the absent type.
The orientation of RS and The relationship between hepatic portal plane and RS plane | up to 30 days after surgery
  the RS plane is an imaginary line drawn along the sulcus and carried across to the base of segment IV and form a "security triangle". Similarly, the hilar plane can also form a triangle in posterior triangle of gallbladder. The areas of these triangles were Compared.

CONTACTS AND LOCATIONS:
Overall Officials: hui hou, master, Study Chair — Second Affiliated Hospital of Anhui Medical University
Locations (1):
- Lei Wang, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: Undecided